CLINICAL TRIAL: NCT02614872
Title: A Proof of Concept (POC) Study, Phase II, Open Label, Randomized, Standard Care - Controlled, Single Center Study Evaluating the Safety and Efficacy of Human, Alpha-1 Antitrypsin (AAT) [GLASSIA®] Treatment in First Lung Transplantation
Brief Title: Study to Evaluate the Safety and Efficacy of Intravenous Glassia® Treatment in Lung Transplantation
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Kamada, Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CT2-LUNG-IV-IL-014
Record Dates: First submitted 2015-11-15; First posted 2015-11-25 (Estimated); Last update posted 2021-09-01 (Actual); Status verified 2019-02

CONDITIONS: Transplantation, Lung Rejection
MeSH Terms: interventions — alpha 1-Antitrypsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- GLASSIA® (Experimental): Glassia® IV treatment additional to Institution standard of care (SOC) for first lung transplant subjects according to Investigator discretion.
  Interventions: Drug: GLASSIA® and Institution standard of care (SOC)
- Institution standard of care (SOC) (No Intervention): Institution standard of care (SOC) for first lung transplant subjects according to Investigator discretion.

INTERVENTIONS:
Drug: GLASSIA® and Institution standard of care (SOC) — Alpha-1 Antitrypsin (AAT) [GLASSIA®] add-on pharmacotherapy and Institution standard of care (SOC)
  Other Names: GLASSIA and Institution standard of care (SOC)
  Arms: GLASSIA®

SUMMARY:
This study evaluates the safety and efficacy of intravenous GLASSIA® treatment in lung transplantation.

DETAILED DESCRIPTION:
There is clinical rationale to advocate the use of AAT(GLASSIA) therapy during episodes of lung inflammation, including acute and chronic rejection. AAT may provide more specifically targeted prevention of pathogenic inflammation, superior to that of general immunosuppressants, with little risk. AAT is the main inhibitor of Neutrophil elastase(NE) in the lower airways and patients with AAT deficiency have low concentrations of the protein in this region of the lung. This explains the proteinase/antiproteinase theory of the development of emphysema in deficient patients in which the amount of elastase released in the lung exceeds the amount of AAT. The net result is persistence of elastase activity leading to lung destruction and the pathological changes of emphysema. Administration of AAT will help to prevent further destruction of the lung architecture and reduce the inflammatory dysregulation that causes pulmonary dysfunction. It is expected that by attacking a specific and previously untreated key component of the pathophysiological cycle of BOS, AAT therapy would decrease the prevalence of BOS in lung transplant recipients and prolong life expectancy of these patients. This will be an open label study in order to ensure safety, in the frame of POC study.

ELIGIBILITY:
Inclusion Criteria:

1. Signed and dated informed consent.
2. Age ≥18 years.
3. Subject is planned to undergo first single or double lung transplant (including heart-lung transplant) as per standard implantation procedure.

Exclusion Criteria:

1. Subject has immunoglobulin A (IgA) deficiency and known anti IgA antibodies.
2. Known history of OR positive serological evidence at the time of screening for hepatitis A virus (HAV), hepatitis B virus (HBV), hepatitis C virus (HCV), Parvovirus B19 (PVB19) or human immunodeficiency virus (HIV) Type 1/2 infection
3. Subjects with a history of severe immediate hypersensitivity reactions, including allergies, anaphylaxis to plasma products or any human proteins of different source.
4. Pregnant or lactating women at entry to study and women of child bearing potential, who are unwilling to agree to continue to use acceptable methods of contraception throughout the study.
5. Presence of psychiatric/ mental disorder or any other medical disorder which might impair the subject's ability to give informed consent or to comply with the requirements of the study protocol.
6. Alcohol abuse or history of alcohol abuse.
7. Illegal drugs.
8. Candidate for organ transplantation other than first lung or heart-lung transplantation
9. Clinically significant bronchial stenosis unresponsive to dilation and/or stenting
10. Participation in another interventional clinical trial within 30 days prior to baseline visit.
11. Inability to attend scheduled clinic visits and/or comply with the study protocol.
12. Any other factor that, in the opinion of the investigator, would prevent the subject from complying with the requirements of the protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2016-07-26 (Actual); Primary Completion 2019-04-11 (Actual); Study Completion 2019-05-07 (Actual)

PRIMARY OUTCOMES:
Incidence of subjects experiencing AEs and/or SAEs | during the study
  Incidence of subjects experiencing causally related AEs and/or SAEs
Incidence and rate of Acute Rejection | per year
  Incidence and rate of Acute Rejection

SECONDARY OUTCOMES:
Annual rate (per subject) of pulmonary infections | per year
  Annual rate (per subject) of pulmonary infections
Incidence of subjects who develop Bronchiolitis Obliterans | during the study
  Incidence of subjects who develop Bronchiolitis Obliterans
Changes in Pulmonary Function Test | Change from baseline and overall effect
  Changes in Pulmonary Function Test

CONTACTS AND LOCATIONS:
Overall Officials: Mordechai Kramer, MD, Principal Investigator — Pulmonary institute, Rabin Medical Center, Israel.
Locations (1):
- Pulmonary Institute - Rabin Medical Center, Petah Tikva, Israel

IPD SHARING:
Plan to Share IPD: No